CLINICAL TRIAL: NCT00008853
Title: Evaluation of Two Type III GBS Polysaccharide-Tetanus Toxoid Conjugate Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: DMID 97-004
Record Dates: First submitted 2001-01-18; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Bacterial Infections; Group B Streptococcus
Keywords: Clinical Evaluation
MeSH Terms: conditions — Bacterial Infections

INTERVENTIONS:
Biological: GBS III-TT-SSI
Biological: GBS III-TT-MPHL

SUMMARY:
The purpose of this study is to test the safety and favorable immune response to an anti-streptococcal vaccine (a vaccine that treats a common bacterial infection) in healthy non-pregnant women.

Group B Streptococcus (GBS) continues to be the single most frequent cause of life-threatening bacterial infection during the first 2 months of life. Further, GBS pregnancy-related morbidity afflicts more than 50,000 women annually in the US. Therefore, active immunization of women is an appealing strategy for the prevention of GBS disease in pregnant women and their infants during the first 3 months of infant life.

DETAILED DESCRIPTION:
In this study 65 healthy, non-pregnant women will receive a single dose of one of two anti-streptococcal vaccinations. Both types of vaccinations are given in upper arm by injection into the muscle. To assess the vaccine effectiveness, patients have blood drawn and examined at weeks 4, 8 and 26, post-vaccination.

ELIGIBILITY:
This information currently is not available.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- AIDS Ctr, New York, New York, United States